CLINICAL TRIAL: NCT03944265
Title: Using Genetics and Shared Decision Making to Improve Lung Cancer Care: A Developmental Study
Brief Title: Genetics and Shared Decision Making in Improving Care for Patients With Stage IVA-C Non-small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18C.584; JT 13163 (Other: JeffTrial Number)
Record Dates: First submitted 2019-04-24; First posted 2019-05-09 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Activating ALK Gene Mutation Negative; Activating EGFR Gene Mutation Negative; Activating ROS1 Gene Mutation Negative; Health Care Provider; Lung Non-Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (treatment decision counseling session) (Experimental): Patients complete a treatment decision counseling session/interview about genetic testing and supportive/palliative care with a qualified member of the research team in-person or via telephone. Health care providers receive a 1-page summary of session results for use in treatment shared decision making at the next office visit.
  Interventions: Other: Counseling; Other: Questionnaire Administration; Other: Medical Chart Review

INTERVENTIONS:
Other: Counseling — Participate in treatment decision counseling session
  Other Names: Counseling Intervention
Other: Questionnaire Administration — Ancillary studies
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review

SUMMARY:
This trial studies the use of genetics and shared decision making in improving care for patients with stage IVA-C non-small cell lung cancer. Developing educational tools may help patients with non-small cell lung cancer to increase patient treatment knowledge, reduce decisional conflict, and promote treatment shared decision making with their health care providers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Use the information on genomic tumor diagnostics, provider treatment recommendations, and patient and provider feedback on the treatment decision making process, which will be used to develop materials and methods to adapt an existing decision counseling program (DCP) for use with patients diagnosed with advanced non-small cell lung carcinoma (NSCLC) as a standard component of clinical care.

SECONDARY OBJECTIVES:

I. Pilot test the adapted DCP in a subset of patients to determine the feasibility of delivering the DCP session.

II. Assess DCP effects on patient treatment knowledge and decisional conflict. III. Assess treatment choice.

OUTLINE:

PHASE I: Use physician input to develop draft treatment education materials and use patient input to adapt an online decision counseling application for use in helping patients clarify treatment preference.

PHASE II: Patients complete a treatment decision counseling session/interview about genetic testing and supportive/palliative care with a qualified member of the research team in-person or via telephone. Health care providers receive a 1-page summary of session results for use in treatment shared decision making at the next office visit.

After completion of study, participants are followed up at 30 and 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with advanced NSCLC (stage IV a-c) that are wild-type for activating genetic alterations (EGFR, ROS 1, and ALK).
* May or may not be candidates for immune checkpoint therapy.
* May have had 1-any number of prior systemic therapy regimens.
* If prior systemic regimen, must have progression disease at time of evaluation.
* Untreated brain metastases permitted.
* Completed pathological analysis of tumor tissue.
* Patients who have exhausted targeting therapy options.
* Can speak and read English.
* All participants must be willing to comply with all study procedures and be available for the duration of the study.
* Providers: Those who treat NSCLC patients as described above.

Exclusion Criteria:

• There are no specific exclusions in this trial for particular medical conditions, comorbidities, or performance status. Any patient deemed appropriate to be considered for evaluation and/or treatment would be appropriate to include in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Development of materials and methods to adapt an existing decision counseling program (DCP) for use with patients diagnosed with advanced non-small cell lung cancer as a standard component of clinical care | Up to 6 weeks
  Results will be reported descriptively. A Decision Counseling Program (DCP) is a tool that allows patients and physicians to engage shared decision making. The DCP will be created based on genetic tumor diagnostics, provider treatment recommendations, and feedback from patients and providers gathered from interviews.

SECONDARY OUTCOMES:
Feasibility of the adapted DCP in a subset of patients: proportion of consenting patients who complete the DCP | Up to 6 weeks
  Results will be reported descriptively. The feasibility endpoint will be the proportion of consenting patients who complete the DCP, about which we will estimate an exact 95% confidence interval by the Clopper-Pearson method.
DCP effects on patient treatment knowledge and decisional conflict | Up to 60 days
  Results will be reported descriptively on pre and post surveys that will be completed by patients Survey is the Decisional Conflict Scale (DCS) Total and subscores have applicable items are a) summed; b) divide by 10; and c) multiplied by 25 Total Score Items 1-10 Score range: 0 [No decisional conflict] to 100 [extremely high decisional conflict].
  Uncertainty Sub score Items 9, 10 Score range: 0 [feels extremely certain about best choice] to 100 [feels extremely uncertain about best choice] Informed Sub score Items 1, 2, 3 Score range: 0 [feels extremely informed] to 100 [feels extremely uninformed].
  Values Clarity Sub score Items 4, 5 Score range: 0 [feels extremely clear about person; a values for benefits and risks/side effects] to 100 [feels extremely unclear about personal value] Support Sub score Items 6, 7, 8 Score range: 0 [feels extremely supported in decision making] to 100 [feels extremely unsupported in decision making]
Treatment choice of patients after receiving counseling | Up to 60 days
  Results will be reported descriptively. Will be collected on pre and post surveys that will be completed by patients. Overall summary statistics will be computed for the patient surveys. Medical records data will be reviewed in order to determine the patient treatment regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Flomenberg, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States